CLINICAL TRIAL: NCT02938416
Title: Comparison of the Functional Recovery and Cytokines Changes Between Isokinetic and Isotonic Training in Patients With Acute Stroke, After Total Hip Replacement or After Total Knee Replacement
Brief Title: The Effect of Isokinetic Strengthening Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Yang Cheng, Visiting Staff Doctor, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CF12251
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Resistance Training; Stroke; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Isokinetic training (Experimental): Ten times, three sets of isokinetic strengthening exercise using 30 degree/sec and 120 degree/sec
  Interventions: Device: Isokinetic strengthening exercise
- Isotonic training (Active Comparator): Ten times, three sets of isotonic strengthening exercise using consistent resistance of 60% of 1-repetition maximum of hip or knee
  Interventions: Device: Isotonic strengthening exercise
- isometric training (Placebo Comparator): home exercise education on isometric quadriceps strengthening on the day of out-patient appointment
  Interventions: Behavioral: isometric strengthening exercise

INTERVENTIONS:
Device: Isokinetic strengthening exercise — Isokinetic strengthening exercise provides muscle training throughout the range of motion of a joint at a pre-set constant speed of angular velocity. It can be performed in an eccentric or concentric way in a controlled manner, and is evidenced to be an effective and safe training method in patients with anterior cruciate ligament reconstruction, burn injury, ankle instability, osteoarthritic knee, and chronic stroke in the past literatures.
  Arms: Isokinetic training
Device: Isotonic strengthening exercise — Isotonic strengthening exercise keeps the tension remained unchanged during the muscle's length changing. As the muscle's force changes via the length-tension relationship during a contraction, an isotonic contraction will keep force constant while velocity changes. There are two types of isotonic contractions: (1) concentric and (2) eccentric. In a concentric contraction, the muscle tension rises to meet the resistance, then remains the same as the muscle shortens. In eccentric, the muscle lengthens due to the resistance being greater than the force the muscle is producing.
  Arms: Isotonic training
Behavioral: isometric strengthening exercise — home exercise education on isometric quadriceps strengthening on the day of out-patient appointment
  Arms: isometric training

SUMMARY:
Our participants will include 40 patients within one month of stroke, 43 patients who received total hip replacement or total knee replacement two to four weeks before. The participants will be randomly assigned to isokinetic, isotonic or isometric training groups. Outcome measures including isometric peak torque of hip/knee at 90 degree of flexion, peak torque of hip/knee at angular velocity of 60 degree/s and 120 degree/s, Short Form 36 (SF-36), the Timed Up and Go test, the Oxford Hip/knee Score, the plasma concentration of hsCRP, and the level of substance P in saliva will be collected at the beginning and 4 weeks after the training program. Statistical significant differences will be determined between the improvement of outcome measures of the isokinetic and the isotonic training groups.

DETAILED DESCRIPTION:
Our participants will include 40 patients within one month of stroke, 43 patients who received total hip replacement or total knee replacement two to four weeks before. The participants will be randomly assigned to isokinetic, isotonic or isometric training groups. Outcome measures including isometric peak torque of hip/knee at 90 degree of flexion, peak torque of hip/knee at angular velocity of 60 degree/s and 120 degree/s, Short Form 36 (SF-36), the Timed Up and Go test, the Oxford Hip/knee Score, the plasma concentration of hsCRP, and the level of substance P in saliva will be collected at the beginning and 4 weeks after the training program. Statistical significant differences will be determined between the

ELIGIBILITY:
Inclusion Criteria:

* within one month of acute stroke
* receive total hip/knee replacement within two to four weeks before

Exclusion Criteria:

* cannot perform from sitting to standing
* Body Mass Index > 30
* Lower limbs fracture history
* Diabetic polyneuropathy
* Cardiopulmonary diseases that impede exercise prescription
* Impaired cognitive function
* Infectious disease during the study period that may cause cytokine changes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2013-01; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Peak torque | 4 weeks
  Isometric peak torque of hip/knee at 90 degree of flexion, peak torque of hip/knee at angular velocity of 60 degree/s and 120 degree/s

SECONDARY OUTCOMES:
Timed Up and Go test | 4 weeks
  stand up from a chair, walk for 3 meters and go back and sit down
Short Form 36 (SF-36) questionnaire | 4 weeks
  Use the 36-item, patient-reported questionnaire to survey the self-perceived health status
Oxford Hip/Knee Score | 4 weeks
  symptoms score during daily activities
The plasma concentration of hsCRP, and the level of substance P in saliva | 4 weeks
  check by drawing blood and test

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Yang Cheng, MD, PhD, Principal Investigator — Department of Physical Medicine and Rehabilitation
Locations (1):
- Department of Physical Medicine and Rehabilitation, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng YY, Chen CH, Wang SP. Isokinetic training of lower extremity during the early stage promote functional restoration in elder patients with disability after Total knee replacement (TKR) - a randomized control trial. BMC Geriatr. 2024 Feb 19;24(1):173. doi: 10.1186/s12877-024-04778-9. PMID 38373934
- [Derived] Cheng YY, Liu CC, Lin SY, Lee CH, Chang ST, Wang SP. Comparison of the Therapeutic Effects Between Isokinetic and Isotonic Strength Training in Patients After Total Knee Replacement: A Prospective, Randomized Controlled Trial. Orthop J Sports Med. 2022 Jun 21;10(6):23259671221105852. doi: 10.1177/23259671221105852. eCollection 2022 Jun. PMID 35757239